CLINICAL TRIAL: NCT06242236
Title: Comparison of Guiding Sedation Level by Respiratory Effort Versus Usual Care in Mechanically Ventilated Patients: A Randomized Controlled Trial (EFFORT-GUIDE Trial 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Phruet Soipetkasem, Critical care medicine, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFORT-GUIDE trial 2; COA No. MURA2023/642 (Other: Ramathibodi hospital)
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: ARDS; Respiratory Effort; Mechanical Ventilation Complication; Sedation
Keywords: Acute respiratory distress syndrome (ARDS); Dynamic transpulmonary pressure swing (Predicted ΔPL); Patient self-inflicted lung injury (P-SILI); Patient ventilator asynchrony (PVA); Respiratory effort
MeSH Terms: conditions — Respiratory Distress Syndrome; Patient-Ventilator Asynchrony

STUDY DESIGN:
Intervention Model Description: The randomized control trial two arms by 1:1 ratio after the participants were recruited.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: respiratory effort guide sedative dosage adjustment. (Active Comparator): Following the enrollment of participants (acute respiratory failure requiring mechanical ventilation which sedation needed), the investigators proceeded to randomize participants into two groups: this intervention group, which employed the optimal respiratory effort parameters to guide the adjustment of sedative levels.
  Interventions: Other: The respiratory effort parameters guide sedative dosage.
- Control group: usual care guide sedative dosage adjustment. (No Intervention): Following the enrollment of participants (acute respiratory failure requiring mechanical ventilation which sedation needed), the investigators proceeded to randomize participants into two groups: this control group, which employed usual care to guide the adjustment of sedative levels.

INTERVENTIONS:
Other: The respiratory effort parameters guide sedative dosage. — The intervention involves the measurement of respiratory effort using P0.1 and Pocc then calculating to dynamic transpulmonary pressure swing (Predicted ΔPL) to adjust sedative drug dosage.
  Other Names: The respiratory effort parameters
  Arms: Intervention group: respiratory effort guide sedative dosage adjustment.

SUMMARY:
The objective of this research is to utilize respiratory effort parameters as a tool to assist in adjusting sedative drug levels for patients undergoing mechanical ventilation in the intensive care unit, in comparison to the conventional usual care approach.

DETAILED DESCRIPTION:
The research investigators conduct daily screening for new participation in the intensive care unit and semi-intensive care unit, selecting individuals based on inclusion and exclusion criteria. In cases where patients require sedative drugs before the research investigators assessment, such as when patients are agitated or have difficulty asynchrony, standard sedative dosages are allowed in emergency rooms and the intensive care unit.

* Informed consent for participation in the research is obtained from direct relatives of participants, accompanied by an explanation of the research procedures, methods, and potential complications. Relatives are required to sign the consent form as the primary decision-makers, considering the participants may be in an altered state of awareness and decision-making capacity.
* Participants meeting the inclusion and exclusion criteria are registered for the research project and assigned a participant identification code. They are divided into two groups: one receiving the intervention involving the measurement of respiratory effort using P0.1 and Pocc then calculating to dynamic transpulmonary pressure swing (Predicted ΔPL) to adjust sedative drugs, and the other, serving as the control group, receives usual care adjustments made by the ward physicians' decision. The randomization process is facilitated by a third party.

The randomization involves creating equally distributed tokens for both groups (1:1 ratio), with the total number (n) representing the population to be included in the study. These tokens are placed in a random box for the randomization process. The basic information of research participants, laboratory, and mechanical ventilator parameters will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged between 18-75 years.
2. Admitted to the critical care and semi-critical care units (ICUs) of the Department of Internal Medicine, Ramathibodi Hospital (ICUs 9IC, 8IK, and 7NW).
3. Patients with acute respiratory failure admitted to the hospital with the following conditions within the first 48 hours:

   * PaO2/FiO2 greater than 150 or
   * PaO2 less than 60 mm Hg or
   * SaO2 less than 90 mm Hg or
   * Work of breathing more than 25 breaths per minute or requiring respiratory muscle assistance
4. Permission obtained from the attending physician.
5. Research participants or their direct relatives must sign informed consent.
6. The research can commence and data can be recorded within 48 hours after the patient has received treatment with the mechanical ventilator.
7. Indicate for receiving sedative drugs during an invasive mechanical ventilator include situations such as when the patient experiences pain or agitation after the placement of the breathing assistance device or when there is patient-ventilator asynchrony.

Exclusion Criteria:

1. Admitted to the hospital or had a history of hospital admission within a month before recruitment.
2. History of cardiovascular or cerebrovascular events within the last 12 months.
3. Allergic to sedative drugs used in the study.
4. Pregnant.
5. Terminal-stage cancer patient, terminal illness-stage of disease who desire palliative care.
6. Active neurological or muscular disorders affecting stability.
7. Brain coma, brain death, or status epilepticus.
8. Severe mental health conditions, including active depression with psychotic features, bipolar disorder, or schizophrenia.
9. Uncontrolled thyroid conditions within a month before recruitment.
10. Uncorrectable patients with severe hypoxemia (P/F ratio less than 150).
11. Patients receiving neuromuscular blocking agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
28 days ventilator-free day | After intubated patients were recruited until successful extubation or dead/failed extubation with in 28 days.
  To compare the number of ventilator-free days at 28 days between the method of measuring respiratory effort using the Dynamic Transpulmonary Pressure Swing (Predicted ΔPL) and P0.1, as opposed to usual care, for adjusting sedative drug dosages in patients with acute respiratory failure requiring mechanical ventilation.

SECONDARY OUTCOMES:
28-day mortality rate | After intubated patients were recruited until alive or dead with in 28 days.
  To compare 28-day mortality rate in patients adjusting sedative drug dosages using the Dynamic Transpulmonary Pressure Swing (Predicted ΔPL) and P0.1 methods compared to usual care.
48 hours the pulmonary mechanics change | After intubated patients were recruited until 48 hours
  To investigate the pulmonary mechanics at 48 hours after sedative drug adjustment using the Dynamic Transpulmonary Pressure Swing (Predicted ΔPL) and P0.1 methods compared to usual care.
The proper respiratory effort level during 48 hours | After intubated patients were recruited until 48 hours
  To determine an appropriate level of respiratory effort and reduce excessive and inadequate effort factors by administering suitable sedative drugs to patients, minimizing lung injury from various causes, with the goal of facilitating the shortest possible duration of mechanical ventilation.
The sedative dosage during 48 hours | After intubated patients were recruited until 48 hours
  To compare the amount of sedative drugs administered to patients within 48 hours after intubation in the intervention group, adjusting drug dosages using the Dynamic Transpulmonary Pressure Swing (Predicted ΔPL) and P0.1 guidance, and the control group, adjusting drug dosages using Usual care guidance. The results will be presented separately for each type of drug, including Propofol infusion rate (mcg/kg/min), midazolam-equivalent infusion rate (mg/hc), fentanyl-equivalent infusion rate (mcg/hd), dexmedetomidine infusion rate (mcg/kg/h).

CONTACTS AND LOCATIONS:
Overall Officials: Pongdhep Theerawit, Assoc. Prof., Study Chair — Critical care medicine Ramathibodi hospital
Locations (1):
- Critical care medicine Ramathibodi hospital, 270 Rama 6 Rd. Phayatai, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
The entire final data results will be shared when the research has been published after a trial period of 2 years.

REFERENCES:
- [Result] Orozco-Levi M, Lloreta J, Minguella J, Serrano S, Broquetas JM, Gea J. Injury of the human diaphragm associated with exertion and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1734-9. doi: 10.1164/ajrccm.164.9.2011150. PMID 11719318
- [Result] Scott A, Wang X, Road JD, Reid WD. Increased injury and intramuscular collagen of the diaphragm in COPD: autopsy observations. Eur Respir J. 2006 Jan;27(1):51-9. doi: 10.1183/09031936.06.00143004. PMID 16387935
- [Result] Moore RL, Binger CA. THE RESPONSE TO RESPIRATORY RESISTANCE : A COMPARISON OF THE EFFECTS PRODUCED BY PARTIAL OBSTRUCTION IN THE INSPIRATORY AND EXPIRATORY PHASES OF RESPIRATION. J Exp Med. 1927 May 31;45(6):1065-80. doi: 10.1084/jem.45.6.1065. PMID 19869306
- [Result] Barach AL, Eckman M. THE EFFECTS OF INHALATION OF HELIUM MIXED WITH OXYGEN ON THE MECHANICS OF RESPIRATION. J Clin Invest. 1936 Jan;15(1):47-61. doi: 10.1172/JCI100758. No abstract available. PMID 16694380
- [Result] Dreyfuss D, Soler P, Basset G, Saumon G. High inflation pressure pulmonary edema. Respective effects of high airway pressure, high tidal volume, and positive end-expiratory pressure. Am Rev Respir Dis. 1988 May;137(5):1159-64. doi: 10.1164/ajrccm/137.5.1159. PMID 3057957
- [Result] Mascheroni D, Kolobow T, Fumagalli R, Moretti MP, Chen V, Buckhold D. Acute respiratory failure following pharmacologically induced hyperventilation: an experimental animal study. Intensive Care Med. 1988;15(1):8-14. doi: 10.1007/BF00255628. PMID 3230208
- [Result] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. The comparison of spontaneous breathing and muscle paralysis in two different severities of experimental lung injury. Crit Care Med. 2013 Feb;41(2):536-45. doi: 10.1097/CCM.0b013e3182711972. PMID 23263584
- [Result] Yoshida T, Torsani V, Gomes S, De Santis RR, Beraldo MA, Costa EL, Tucci MR, Zin WA, Kavanagh BP, Amato MB. Spontaneous effort causes occult pendelluft during mechanical ventilation. Am J Respir Crit Care Med. 2013 Dec 15;188(12):1420-7. doi: 10.1164/rccm.201303-0539OC. PMID 24199628
- [Result] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Result] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Result] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Result] Taran Z, Namadian M, Faghihzadeh S, Naghibi T. The Effect of Sedation Protocol Using Richmond Agitation-Sedation Scale (RASS) on Some Clinical Outcomes of Mechanically Ventilated Patients in Intensive Care Units: a Randomized Clinical Trial. J Caring Sci. 2019 Dec 1;8(4):199-206. doi: 10.15171/jcs.2019.028. eCollection 2019 Dec. PMID 31915621
- [Result] Karamchandani K, Rewari V, Trikha A, Batra RK. Bispectral index correlates well with Richmond agitation sedation scale in mechanically ventilated critically ill patients. J Anesth. 2010 Jun;24(3):394-8. doi: 10.1007/s00540-010-0915-4. Epub 2010 Mar 12. PMID 20225074
- [Result] Dzierba AL, Khalil AM, Derry KL, Madahar P, Beitler JR. Discordance Between Respiratory Drive and Sedation Depth in Critically Ill Patients Receiving Mechanical Ventilation. Crit Care Med. 2021 Dec 1;49(12):2090-2101. doi: 10.1097/CCM.0000000000005113. PMID 34115638
- [Result] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Result] Bertoni M, Spadaro S, Goligher EC. Monitoring Patient Respiratory Effort During Mechanical Ventilation: Lung and Diaphragm-Protective Ventilation. Crit Care. 2020 Mar 24;24(1):106. doi: 10.1186/s13054-020-2777-y. PMID 32204729

DOCUMENTS (1):
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT06242236/ICF_000.pdf